CLINICAL TRIAL: NCT05212207
Title: Forecasting and Preventing Post-Bariatric Hypoglycaemia (Work Package 1)
Brief Title: Forecasting and Preventing Post-Bariatric Hypoglycaemia WP 1
Acronym: PBH Forecast
Status: Completed | Type: Observational
Sponsor: Lia Bally (Other)
Collaborators: University of Padova (Other)
Responsible Party: Sponsor-Investigator, Lia Bally, Head of Nutrition, Metabolism and Obesity and Head of Research, Insel Gruppe AG, University Hospital Bern
Organization: Insel Gruppe AG, University Hospital Bern (Other)
Other Study IDs: PBH Forecast (WP 1)
Record Dates: First submitted 2022-01-14; First posted 2022-01-28 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Post-bariatric Hypoglycaemia; Roux-en-Y Gastric Bypass
Keywords: Continuous Glucose Monitoring
MeSH Terms: interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PBH
  Interventions: Other: CGM, smartwatch, and electronic diary

INTERVENTIONS:
Other: CGM, smartwatch, and electronic diary — Participants wear a CGM and a smartwatch while keeping an electronic diary with information such as meals, sleep, and activity.

SUMMARY:
The overall aim of this study is to prevent hypoglycemic events in patients with hypoglycemia after a meal and to develop a sustainable hypoglycemia correction strategy.

DETAILED DESCRIPTION:
Obesity is a major global public health concern, for which the most effective therapy is bariatric surgery. Beyond weight loss, bariatric surgery exerts powerful effects on glucose metabolism, achieving complete type 2 diabetes remission in up to 70% of cases. An exaggeration of these effects, however, can result in an increasingly recognized metabolic complication known as postprandial hyperinsulinaemic hypoglycaemia or post-bariatric hypoglycaemia (PBH). The condition manifests 1-3 years after surgery with meal-induced hypoglycaemic episodes. Emerging data suggests that PBH is more frequent than previously thought and affects approximately 30% of postoperative patients, more commonly after gastric bypass than sleeve gastrectomy. Of note, asymptomatic PBH is common, as shown in studies using continuous glucose monitoring (CGM). It is known from extensive research in people with diabetes that recurrent episodes of hypoglycaemia impair counter regulatory defences against subsequent events, predisposing patients to severe hypoglycaemia.

Despite the increasing prevalence of PBH, clinical implications in this population are still unclear. Anecdotal evidence from patients with PBH suggests a high burden for these patients due to the recurrent hypoglycaemias with possibly debilitating consequences. It is well established that even mild hypoglycaemia (plasma glucose of 3.4 mmol/L) in diabetic and non-diabetic patients impairs various cognitive domains. Of note, some of the cognitive functions remain impaired for up to 75 min, even when the hypoglycaemia is corrected. Further concerns exist from observational studies showing associations between PBH during pregnancy and poor foetal growth.

Thus, it is important to timely detect and treat hypoglycaemia with an intervention that allows quick recovery of glycaemia to a safe level, thereby alleviating symptoms and eliminating the risk of potentially hazardous sequelae. Recently, CGM devices have become standard tools for glucose monitoring in patients with diabetes. CGM allows measuring glucose levels every 5 min and the continuous access to real-time data offering several approaches for the prediction of glucose levels or associated events. Such solutions empower patients to take proactive decisions before reaching critical glucose levels. Apart from glucose levels, meal information, physical activity or other physiological parameters may augment prediction performance of hypoglycaemic events. While most engineering work focuses on the prediction of hypoglycaemia in the diabetic population, only preliminary work has been done in the PBH population.

Given the potentially hazardous consequences of hypoglycaemia, development of hypoglycaemia management strategies to adequately predict and treat critical blood glucose levels in the PBH population are urgently needed. Such strategies have to significantly lower the burden of PBH and increase patient safety.

The overall aim or this study is to prevent hypoglycaemic events in patients with PBH and to develop a sustainable hypoglycaemia correction strategy.

The primary objective of WP 1 is to develop a hypoglycaemia prediction model based on sensor glucose data. Furthermore, the investigators will try to improve the prediction by including further data streams such as information about meal intake, heart rate and activity data.

ELIGIBILITY:
Inclusion Criteria:

* Post-bariatric surgery patients (Roux-en-Y gastric bypass) with PBH, defined as postprandial plasma or sensor glucose <3.0 mmol/L according to the International Hypoglycaemia Study Group and exclusion of other causes of hypoglycaemia
* Age ≥18 years

Exclusion Criteria:

* Inability to give informed consent as documented by signature
* Pregnant or lactating women
* Inability or contraindications to undergo the investigated intervention
* Drugs interfering with blood glucose (e.g. SGLT-2 inhibitors, acarbose) during the time of investigation
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of post-bariatric patients with PBH.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
Precision (fraction of correct alarms over the total number of raised alarms) and recall (fraction of correctly predicted hypoglycaemic events over the total number of episodes) | 10 days
  Selecting the best performing hypoglycaemia prediction

SECONDARY OUTCOMES:
False alarms | 10 days
  Daily number of false alarms triggered by the algorithms (FP-per-day)
Time anticipation | 10 days
  Time anticipation between the hypoglycaemic alarms raised by the model and the hypoglycaemic episode

CONTACTS AND LOCATIONS:
Overall Officials: Lia Bally, Prof. Dr. med. et phil., Principal Investigator — Department of Diabetes, Endocrinology, Nutritional Medicine and Metabolism, lnselspital, Bern University Hospital, University of Bern
Locations (1):
- Department of Diabetes, Endocrinology, Nutritional Medicine and Metabolism (UDEM), Inselspital, Bern University Hospital, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be available to other researchers.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After study completion, 10 years
Access Criteria: After written inquiry and approval by the principal investigator.